CLINICAL TRIAL: NCT04969601
Title: Anti-Covid-19 Vaccine Protection in Immunocompromised Children (1 to 15 Years Old) With Acute Leukemia and Their Siblings (≥12 Years Old). Phase I-II Trial Evaluating Post-vaccine Safety and Humoral and Cellular Immunogenicity.
Brief Title: Anti-Covid-19 Vaccine in Children With Acute Leukemia and Their Siblings
Acronym: PACIFIC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APHP210639
Record Dates: First submitted 2021-07-19; First posted 2021-07-20 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Acute Leukemia; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — BNT162 Vaccine

STUDY DESIGN:
Intervention Model Description: Dose finding, stratified on the age group (≥1-<2 years, ≥2-<5 years, ≥5-<12 years)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti Covid with COMIRNATY® (BNT162b2) vaccine (Experimental): Two injections of COMIRNATY® (BNT162b2) vaccine 21-28 days apart
  Interventions: Biological: vaccine COMIRNATY® (BNT162b2)

INTERVENTIONS:
Biological: vaccine COMIRNATY® (BNT162b2) — two injections of COMIRNATY® (BNT162b2) vaccine 21-28 days apart, of either 10, 20, 30 µg of vaccine, depending on the observed responses of previous children

SUMMARY:
Mortality in case of SARS-CoV-2 infection (Covid-19) during acute leukemia (AL) treatment is around 30%, i.e. more than 10 times the one of general population. Severe forms are reported in children receiving chemotherapy for AL. However, the main risk, largely underestimated, is related to delay in chemotherapy administration in case of infection, leading to an increased risk of relapse. Therefore, it is justified to propose an anti-Covid-19 vaccination to these patients. Vaccination of siblings also seems necessary given the uncertainty regarding vaccine response in children with AL and given that household is the main source of contamination. The messenger ribonucleic acid (mRNA) vaccine COMIRNATY® (BNT162b2) is already approved by health authorities for individuals older than 12. In immunocompromised children with AL, safety and efficacy data are unknown. The benefit/risk balance encourages to use the vaccine without health authority approval in children aged 1 to 15 with AL. Regarding household, parents are vaccinated for several months as standard of care, but vaccination will be proposed to siblings aged 5 to 15 years old in this protocol.

The primary objective of this study is to evaluate safety and immunogenicity of COMIRNATY® (BNT162b2) vaccine (two injections 21-28 days apart) in children with acute leukemia (1 to 15 years old) and their siblings (5 to 15 years old).

A secondary objective of the study is to compare the quality of humoral and cellular vaccine responses in children with AL and healthy children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to 15 years old :

  * With acute lymphoblastic leukemia undergoing chemotherapy (at least 2 weeks from the last injection of PEG-asparaginase) or for whom the last chemotherapy is less than or equal to 12 months
  * OR With acute myeloid leukemia within 12 months from the end of treatment
* Healthy siblings aged 5 to 15 years old living in the same household than the child with AL more than 50% of the time
* Informed consent from parents
* Patient affiliated to health insurance
* For women of childbearing age :

  * A negative blood test at the inclusion visit
  * AND use of an effective contraceptive method at least at least 4 weeks prior to vaccination and until at least 12 weeks after the last vaccination

Exclusion Criteria:

* Documented SARS-CoV-2 infection ongoing or that occurred less than 2 months ago
* Known clinical allergy to polyethylene glycol (PEG)
* Platelet <50 Giga(G) G/L or neutrophils <0.5 G/L at time of vaccination
* Vaccination apart from influenza virus within 4 weeks from the 1st injection or planning to receive an approved vaccine 4 weeks after the last injection
* Vaccination against influenza virus within 14 days before first injection
* Any hemorrhagic trouble considered as a contraindication to intramuscular injection
* History of severe adverse event after a vaccine administration including anaphylaxis and associated symptoms such as rash, respiratory issues, angioedema and abdominal pain, or history of allergic reaction that could be exacerbated by a vaccine component
* Participant vaccinated against tuberculosis within the past year
* Participant ill or febrile (body temperature ≥38°C) in the previous 72 hours with symptoms suggesting the presence of COVID-19.
* Allergy to any component of the vaccine or history of severe allergy (anaphylactic type)
* Treatment received for Covid-19 infection (60 days prior to 1st injection).
* Known HIV, HCV or HBV infection.
* Use of experimental Ig, experimental monoclonal antibodies or convalescent anti-covid-19 serum within 90 days prior to study entry
* Pregnant, breast-feeding or positive pregnancy test at inclusion visit.
* Participation in a vaccination trial
* Participation in other research without investigator's consent research within 4 weeks prior to the inclusion visit and for the duration of the trial

Translated with DeepL.com (free version)

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | within 7 days from first dose
  Dose limiting toxicity (DLT) defined by the presence within 7 days following vaccine injection of a grade ≥3 adverse event related to the vaccine. They are derived from CTCAE v5.0 and FDA guide " Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials ".
  Any other unexpected grade 3-4 clinical adverse event according to CTCAE v5.0 related to vaccination.
  A committee of critical events and DLTs surveillance will validate if declared grade 3-4 serious adverse events are related to vaccine.
co-primary endpoint: anti-Spike Immunoglobulin G (IgG) titer >= 260 BAU/mL | at 1 month from second dose
  Quantitative detection of anti-spike antibodies by chemiluminescence technique

SECONDARY OUTCOMES:
Anti-Spike IgG levels | between 21 and 28 days from first dose
Anti-Spike IgG levels | at 6 months from first dose
Anti-Spike IgG levels | at 12 months from the 1st dose
Anti-nucleocapsid IgG levels | between 21 and 28 days from the first dose
Anti-nucleocapsid IgG levels | 6 months from the first dose
Anti-nucleocapsid IgG levels | 12 months from the first dose
Neutralization ability of anti-Spike IgG (in case of anti-Spike IgG detection) | at 2 months from the first injection
Neutralization ability of anti-Spike IgG (in case of anti-Spike IgG detection) | at 6 months from the first injection
Neutralization ability of anti-Spike IgG (in case of anti-Spike IgG detection) | at 12 months from the first injection
Anti-SARS-CoV-2 T cell specific response (Elispot) | at 2 months after the first injection
Anti-SARS-CoV-2 T cell specific response (Elispot) | at 6 months after the first injection
Anti-SARS-CoV-2 T cell specific response (Elispot) | at 12 months after the first injection
Positivity of SARS-CoV-2 polymerase chain reaction (PCR) in nasopharynx | at 8 days
  Positivity of SARS-CoV-2 PCR in nasopharynx in case of infection
Positivity of SARS-CoV-2 PCR in nasopharynx | at 15 days
  Positivity of SARS-CoV-2 PCR in nasopharynx in case of infection
Positivity of SARS-CoV-2 PCR in nasopharynx | at 28 days from infection
  Positivity of SARS-CoV-2 PCR in nasopharynx in case of infection
Rate of symptomatic SARS-CoV-2 infections | within 12 months after vaccination
  Symptomatic SARS-CoV-2 infections will be defined by the presence of at least one symptom amongst fever, dyspnea, cough, chest pain, anosmia, ageusia, diarrhea or vomiting, AND a positive SARS-CoV-2 PCR,
Genotype of the SARS-CoV-2 variant in case of infection | within 12 months after vaccination
Time between chemotherapy planned date and effective date in case of infection | within 12 months after vaccination
Covid19 World Health Organization (WHO) progression scale | within 12 months after vaccination
  Covid19 WHO scale in 10 items in case of infection Uninfected; non viral RNA detected: 0 Asymptomatic; viral RNA detected: 1 Symptomatic; Independent: 2 Symptomatic; Assistance needed: 3 Hospitalized; No oxygen therapy: 4 Hospitalized; oxygen by mask or nasal prongs: 5 Hospitalized; oxygen by non-invasive ventilation (NIV) or High flow: 6 Intubation and Mechanical ventilation, pO2/Fraction of inspired oxygen (FIO2)>=150 OR saturation by pulse oximetry (SpO2) SpO2/FIO2>=200: 7 Mechanical ventilation, (pO2/FIO2<150 OR SpO2/FIO2<200) OR vasopressors (norepinephrine >0.3 microg/kg/min): 8 Mechanical ventilation, pO2/FIO2<150 AND vasopressors (norepinephrine >0.3 microg/kg/min), OR Dialysis OR extracorporeal membrane oxygenation (ECMO): 9 Dead: 10
Incidence of SARS-CoV-2 of the household (contact cases) | within 12 months after vaccination
  In case of infection in a vaccinated child

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Armand Trousseau, Paris
  - Hôpital Robert Debré, Paris

IPD SHARING:
Plan to Share IPD: Undecided